CLINICAL TRIAL: NCT04444960
Title: Prospective Registry of the Intracoronary Physiology and Imaging-guided Precision Therapy in Complex High-risk Patients
Brief Title: Precision Therapy in Complex High-risk Coronary Artery Disease
Acronym: PTCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2019-014
Record Dates: First submitted 2020-06-21; First posted 2020-06-24 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intracoronary physiology and imaging-guided group
  Interventions: Procedure: percutaneous coronary intervention
- Angiography-guided group
  Interventions: Procedure: percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — Intracoronary physiology and imaging-guided intervention strategy versus angiography-guided intervention strategy for complex high-risk coronary heart disease patients

SUMMARY:
This is a prospective registry to enroll complex high-risk coronary heart disease patients.

The purpose of this study is to compare intracoronary physiology and imaging-guided intervention strategy and angiography-guided intervention strategy for clinical outcomes and health economics.

ELIGIBILITY:
Inclusion Criteria:

* Bifurcation lesions with branch diameter ≥2.5mm;
* Chronic complete occlusion (occlusion duration ≥3 months);
* Left main disease;
* Long lesions (≥38mm);
* Multi-vessel percutaneous coronary intervention (simultaneous treatment of ≥2 epicardial vessels during one operation);
* Multi-stent implantation (≥3 stents);
* In-stent restenosis;
* Moderate to severe calcification on radiography;
* Intermediate lesion;
* Thrombotic lesions;
* Creatinine clearance rate < 60ml/min) or on dialysis ;
* Left ventricular ejection fraction <40% ；
* History of cerebral hemorrhage or massive hemorrhage of gastrointestinal tract.

Exclusion Criteria:

* Informed consent cannot be obtained;
* Life expectancy < 1 year.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Coronary heart disease patients with complicated clinical conditions and/or complex coronary lesions.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Composite ischemic events | 24 months
  Composite ischemic event is defined as the composite of cardiac death, stent thrombosis, nonfatal myocardial infarction or ischemic driven revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Huang, phD, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China